CLINICAL TRIAL: NCT06984133
Title: Evaluating the Effectiveness of a Structured Educational Program on Glycemic Control in Adolescents With Type 1 Diabetes: A Randomized Controlled Trial
Brief Title: Structured Education Program and Glycemic Control in Adolescents With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA HM-2025-02
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes (T1D); Type 1 Diabetes Mellitus (T1DM)
Keywords: Kuwait; Glycemic control; Type 1 diabetes; Carbohydrate counting; Arab adolescents; Structured education; Adolescents; Diabetes education program; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigators and data analysts will be masked to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Participants will receive usual care at their treating hospitals.
- Intervention arm (Experimental): Participants will attend a structured education program over 4 days and a refresher course after 6 months.
  Interventions: Behavioral: Structured education program

INTERVENTIONS:
Behavioral: Structured education program — A structured group educational program culturally adapted from a UK model for adolescents with type 1 diabetes. The program aims to empower adolescents by providing knowledge and tools needed for effective diabetes management.
  It is delivered by dietitians, diabetes educators, and a pediatric endocrinologist in small groups. The curriculum targets both caregivers and adolescents: the first day is for parents and covers diabetes basics, management of hypoglycemia and hyperglycemia, insulin dosing, sick day management, and exercise considerations. The following three days focus on adolescents and include interactive sessions on the role of food in diabetes management, the effect of different nutrients on blood glucose levels, carbohydrate sources, reading food labels, advanced carbohydrate counting, and insulin dose adjustment.
  Arms: Intervention arm

SUMMARY:
Type 1 diabetes is becoming more common in Kuwaiti and Arab adolescents. Many young people with this condition struggle to keep their blood glucose levels under control, which can lead to diabetes-related complications and affect their quality of life.

The goal of this clinical trial is to evaluate the effectiveness of a structured educational program on glycemic control among Arab adolescents with type 1 diabetes aged 11 to 14 years.

Participants will be randomly assigned to one of two groups. The intervention group will receive the structured education program, and the control group will continue with standard care.

All participants will undergo assessments that include:

* collecting demographic and diabetes management data
* measuring weight and height
* measuring HbA1c levels and lipid profile
* filling out questionnaires on quality of life, carbohydrate and insulin dosing knowledge, physical activity
* collecting dietary intake
* providing AGP report

Participants in the intervention group will additionally be required to:

* attend the program for 4 consecutive days, one day for parents and three days for children
* fill out 3-day food diary records during the program
* attend a refresher course after 6 months

Participants in the control group will have the opportunity to participate in the program after approximately six months.

ELIGIBILITY:
Inclusion Criteria:

* Arab adolescents
* Males and females aged 11 to 14 years.
* Have been diagnosed with type 1 diabetes for at least 6 months.
* Wearing a continuous glucose monitor (CGM).
* Individuals and their parents must be able to join the entire duration of the study.
* Individuals and their parents must voluntarily provide consent and assent.

Exclusion Criteria:

* Presence of learning disabilities or any known psychological issues.
* Attendance at any diabetes education or carbohydrate counting programs within the six months preceding the study.

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2025-05-18 (Estimated); Primary Completion 2028-05-18 (Estimated); Study Completion 2028-05-18 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c Levels | Baseline and 6 months
  Change in HbA1c Levels from baseline to 6 months
Change in %Time In Range (%TIR) | Baseline and 6 months
  Change in %TIR from baseline to 6 months

SECONDARY OUTCOMES:
Change in Carbohydrate Counting and Insulin Adjustment Knowledge Scores | Baseline and 6 months
  Change in Carbohydrate Counting and Insulin Adjustment Knowledge Scores from baseline to 6 months
Change in Diabetes-Specific Quality of Life Scores | Baseline and 6 months
  Change in Diabetes-Specific Quality of Life Scores from baseline to 6 months, will be assessed using the validated Arabic version of the Pediatric Quality of Life Inventory 3.0 Diabetes Module (PedsQL DM).
Change in Hypoglycemia Frequency | Baseline and 6 months
  This will be assessed by:
  a) the percentage of time blood glucose levels are below the target range (%TBR), and b) parent-reported episodes requiring treatment such as glucagon administration.
Change in Diabetes-Related Hospitalizations | Baseline and 6 months
  Frequency of hospital admissions for diabetic ketoacidosis or hypoglycemia, reported by parents, within a month prior the assessment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa Al Ozairi, MD, Study Director — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Sharq, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided